CLINICAL TRIAL: NCT03465371
Title: CSC OnDemand: An Innovative Online Learning Platform for Implementing Coordinated Specialty Care
Acronym: CSCPII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Collaborators: Dartmouth College (Other); University of Maryland (Other); New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4R44MH111283-02 (NIH)
Record Dates: First submitted 2018-02-20; First posted 2018-03-14 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A 3-arm randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OnDemand Training Intervention (Experimental): Participants receiving the OnDemand Training Intervention
  Interventions: Other: CSC OnDemand Training Intervention
- InPerson Intervention (Active Comparator): Participants receiving the InPerson Intervention
  Interventions: Other: InPerson Intervention
- Virtual InPerson Intervention (Active Comparator): Participants receiving the Virtual InPerson Intervention (the InPerson training via Zoom)
  Interventions: Other: Virtual InPerson Intervention

INTERVENTIONS:
Other: CSC OnDemand Training Intervention — Level 1: Readiness
  Online readiness tool
  Level 2: Core Knowledge
  Week 1-self-paced core curriculum, totaling 8 hours of instruction
  Level 3: Going Deeper
  Week 2-instructor-led, role-specific, and advanced topics, totaling 12 hours of instruction
  Level 4: Sustainability
  9 months of online community of practice support; a discussion forum; open office hours with experts; multisite case conferencing; access to online materials
  Arms: OnDemand Training Intervention
Other: InPerson Intervention — Level 1: Readiness
  Telephone conversations with program leaders to determine structures, roles, staffing, recruitment
  Level 2: Core Knowledge
  1 day of in-person training on FEP basics and CSC components
  Level 3: Going Deeper
  1.5 days of in-person training on how the team works, followed by breakout sessions by role
  Level 4: Sustainability
  9 months of monthly implementation coaching calls with team leads; monthly telephone case conferences; monthly care coordination calls split out by role
  Arms: InPerson Intervention
Other: Virtual InPerson Intervention — Level 1: Readiness
  Telephone conversations with program leaders to determine structures, roles, staffing, recruitment
  Level 2: Core Knowledge
  1 day of virtual (via Zoom) in-person training on FEP basics and CSC components
  Level 3: Going Deeper
  1.5 days of virtual (via Zoom) in-person training on how the team works, followed by breakout sessions by role
  Level 4: Sustainability
  9 months of monthly implementation coaching calls with team leads; monthly telephone case conferences; monthly care coordination calls split out by role
  Arms: Virtual InPerson Intervention

SUMMARY:
In response to the growing need for training on interventions to address first episode psychosis, the Center for Social Innovation (C4) partnered with experts in Coordinated Specialty Care (CSC) to develop and test CSC OnDemand: An Innovative Online Learning Platform for Implementing Coordinated Specialty Care. The product builds on the findings of the Recovery After an Initial Schizophrenia Episode (RAISE) studies, funded by the National Institute of Mental Health (NIMH). RAISE examined team-based models of care for people early in the course of schizophrenia. Through a Fast Track Small Business Innovation Research (SBIR) grant, investigators will prototype, test, refine, and evaluate the impact of CSC OnDemand.

DETAILED DESCRIPTION:
Building on existing resources and the expertise of our faculty and advisors, the investigators developed CSC OnDemand, a multifaceted online learning product that includes four levels: 1) an online readiness tool and CSC Learning Hub; 2) dynamic multimedia core curriculum on first episode psychosis and CSC; 3) live faculty-led online courses; and 4) ongoing support, including an online community of practice to support peer-to-peer learning.

During Phases I and II of this Fast Track SBIR, the investigators prototyped, pilot tested, built out, and evaluated the product through a cluster randomized study comparing it with InPerson training (and due to the global pandemic, a "virtual" in person training, using Zoom to train with the same curriculum as in-person, creating (unexpectedly) three study arms).

Phase I built a robust prototype of the online platform and tested it with 16 providers from three sites. This phase explored feasibility, acceptability, and preliminary effectiveness of the product, and examined which components of the online platform providers found most useful.

Based on our findings from Phase I, the investigators refined and fully built out the product to test in a larger randomized trial. Phase II used a cluster randomized non-inferiority design to assess if OnDemand training (n = 20 sites) was comparable to InPerson training (n = 10 sites). Using a mixed-methods approach, the investigators examined provider (n enrolled was 239; after attrition 206) outcomes (satisfaction; knowledge gains/retention; attitudes toward shared decision making) and client (n = 110) outcomes (work/school participation; engagement in CSC services; inpatient psychiatric hospitalizations).

The study was guided by the following specific aims:

Phase II AIM 1: To refine, expand, and finalize CSC OnDemand based on Phase I findings.

AIM 2: To examine the differences in outcomes of OnDemand training intervention as compared to the InPerson and Virtual In Person interventions as it related to CSC providers knowledge and shared decision making (SDM). Hypothesis: Providers in the OnDemand condition will achieve increases in knowledge, SDM and satisfaction at post training and nine months that will be no more than .5 standard deviations less than the InPerson or Virtual InPerson condition.

AIM 3: To determine if the OnDemand training intervention is as successful as the InPerson or Virtual InPerson training in increasing participation in work or school, improving engagement in treatment, and decreasing relapse rates for participating clients. Hypothesis: Clients being served by the providers in the OnDemand condition will have work/school participation rates, levels of engagement and rates of hospitalization nine months after admission that are no more than 10 percent higher (hospitalization) or lower (work/school, engagement) than clients served by providers in the InPerson or Virtual InPerson condition.

ELIGIBILITY:
Inclusion Criteria:

Agencies will need to provide:

* direct care to individuals with early psychosis;
* administrative-level support for training and use of the CSC model;
* an entire treatment team that is willing to participate in this team-based intervention;
* contact information for direct service staff;
* support for the study, including a staff person to serve as a liaison to work with the research team;
* access to the Internet during the intervention period; and
* a willingness to provide data and participate in the evaluation.

Exclusion Criteria:

* Teams should not have previously received CSC training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Provider-level: Success in increasing CSC providers knowledge of CSC | Up to 9 months
  CSC knowledge will be assessed with a 50-item, complex, multiple-choice test (25 common across disciplines, 25 discipline-specific), which will be created in conjunction with the intervention modules and will be piloted in Phase I. The outcome will be the percentage of correct responses.
Provider-level: Success in increasing CSC providers shared decision making | Up to 9 months
  Shared Decision Making Questionnaire-physician version (SDM-Q-Doc) is a standardized brief instrument (9 items) for assessing SDM in clinical encounters. SDM-Q-Doc was developed for physicians, but has been adapted to all healthcare professionals. The instrument consists of 9 statements rated on a 6-point scale from "completely disagree" (0) to "completely agree" (5). The items are summed to create a total score.

SECONDARY OUTCOMES:
Client-level: Work/School Participation | Up to 9 months
  Work/school participation (any work or school participation in the prior three months) will be assessed by the team at baseline, three months, six months, and nine months.
Client-level: Engagement | Up to 9 months
  The time to last mental health visit will be truncated at the nine-month point, so the investigators will use a binary indicator (yes/no) of continued treatment participation at nine months.
Client-level: Psychiatric Hospitalization | Up to 9 months
  The investigators will use a binary indicator of whether the client has been hospitalized in the first nine months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ferreira, PhD, Principal Investigator — C4 Innovations
Locations (1):
- Center for Social Innovation, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes